CLINICAL TRIAL: NCT07184203
Title: Comparative Clinicomycologic and Dermoscopic Study Between Daily and Pulse Therapy of Oral Itraconazole in Tinea Capitis in Children
Brief Title: Comparison Between Continuous and Pulse Itraconazole in Tinea Capitis in Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Marina Aioub, general practitioner, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0108853
Record Dates: First submitted 2025-09-14; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-02

CONDITIONS: Tinea Capitis
MeSH Terms: conditions — Tinea Capitis | interventions — Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A will receive itraconazole continuous daily regimen (Active Comparator)
  Interventions: Drug: Itraconazole (ITZ)
- Group B will receive itraconazole pulse regimen (Active Comparator)
  Interventions: Drug: Itraconazole (ITZ)

INTERVENTIONS:
Drug: Itraconazole (ITZ) — therapy for tinea capitis orally

SUMMARY:
A study to compare the efficacy of daily therapy versus pulse therapy of oral itraconazole in the treatment of tinea capitis in children based on clinical, mycological and dermoscopic evaluation.

ELIGIBILITY:
Inclusion Criteria:

• Tinea capitis patients with ages ranging from 5 to 18 year

Exclusion Criteria:

* Patients with contraindications to itraconazole
* Patients with associated scalp disease.
* Patients weighing less than 20 Kg.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-03-09 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
improvement of tinea capitis | 3 months
  cure of tinea capitis

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No